CLINICAL TRIAL: NCT04462731
Title: Postoperative Pain After One-visit Root Canal Treatment on Teeth With Vital Pulps: Comparison of Two Different Root Filling Techniques
Brief Title: Post-endodontic Pain Survey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ya-Hsin Yu, DDS, MS (Other)
Responsible Party: Sponsor-Investigator, Ya-Hsin Yu, DDS, MS, Principal Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 825494
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain; Endodontic Disease; Obturation
Keywords: Postoperative Pain; Bioceramic; Root canal filling
MeSH Terms: conditions — Pain, Postoperative; Dental Pulp Diseases; Bites and Stings | interventions — Serum Bactericidal Test

STUDY DESIGN:
Intervention Model Description: Non-surgical root canal treatment:
  All teeth were isolated with a rubber dam during root canal treatment. The procedures were performed under a microscope (OPMI Pico; Carl Zeiss, Gottingen, Germany). After access, location of canals, and determination of working length (WL) with Root ZX II apex locator (J Morita, Kyoto, Japan), the canals were instrumented using various .04 taper rotary NiTi instruments to a minimum apical size of 35. 4% NaOCl was used as the main irrigant. 17% EDTA was used as the final irrigant. Passive ultrasonic irrigation with size 20 Acteon tip inserted 2mm short of WL was performed with both 4% NaOCl and 17% EDTA for 10 seconds in each canal. After final irrigation, the canals were dried with paper points. The master gutta-percha cone fit was verified with periapical radiographs before filling the tooth.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obturation technique: WVT (Experimental): Warm vertical compaction technique (WVT): Teeth filled with AH Plus Jet Root Canal Sealer were filled with .04 taper gutta-percha points by WVT. The sealer was introduced with the master cone. The depth of heated plugger was within 3-5 mm of WL in the WVT group, and the remaining canal space was backfilled with additional sealer and thermoplasticized gutta-percha.
  Interventions: Procedure: Non-surgical root canal treatment filled with WVT
- Obturation technique: SBT (Active Comparator): Sealer-based filling technique (SBT): Teeth filled with SBT were obturated with EndoSequence BC Sealer by injecting the sealer into the coronal third of each canal. Size 30 Lentulo spiral coated with additional sealer was introduced 3 mm short of WL depth at 300rpm. Bioceramic coated gutta-percha was dipped in BC sealer and introduced into the canal to WL. A heated plugger was used to sear the gutta-percha point at each orifice.
  Interventions: Procedure: Non-surgical root canal treatment filled with SBT

INTERVENTIONS:
Procedure: Non-surgical root canal treatment filled with WVT — All eligible teeth were isolated with a rubber dam during root canal treatment. The procedures were performed under a microscope (OPMI Pico; Carl Zeiss, Gottingen, Germany). After access, location of canals, and determination of working length (WL) with Root ZX II apex locator (J Morita, Kyoto, Japan), the canals were instrumented using various .04 taper rotary NiTi instruments to a minimum apical size of 35. 4% Sodium hypochlorite was used as the main irrigant with a 31-gauge needle. 17% EDTA was used as the final irrigant. Passive ultrasonic irrigation with size 20 Acteon tip inserted 2mm short of WL was performed with both 4% sodium hypochlorite and 17% EDTA for 10 seconds in each canal. After final irrigation, the canals were dried with paper points. The master gutta-percha cone fit was verified with periapical radiographs before filling the tooth. WVT was used to fill the tooth when the months were January, March, May, July, September, and November.
  Arms: Obturation technique: WVT
Procedure: Non-surgical root canal treatment filled with SBT — All eligible teeth were isolated with a rubber dam during root canal treatment. The procedures were performed under a microscope (OPMI Pico; Carl Zeiss, Gottingen, Germany). After access, location of canals, and determination of working length (WL) with Root ZX II apex locator (J Morita, Kyoto, Japan), the canals were instrumented using various .04 taper rotary NiTi instruments to a minimum apical size of 35. 4% Sodium hypochlorite was used as the main irrigant with a 31-gauge needle. 17% EDTA was used as the final irrigant. Passive ultrasonic irrigation with size 20 Acteon tip inserted 2mm short of WL was performed with both 4% sodium hypochlorite and 17% EDTA for 10 seconds in each canal. After final irrigation, the canals were dried with paper points. The master gutta-percha cone fit was verified with periapical radiographs before filling the tooth. SBT was used to fill the tooth when the months were February, April, June, August, October, and December.
  Arms: Obturation technique: SBT

SUMMARY:
As part of root canal treatment, canals should be sealed to prevent further contaminations. There are multiple accepted techniques to fill-obturate canals. In the past, different obturation techniques have been compared. The most current technique used, a single cone with bioceramic sealer, has not been compared. This clinical investigation will compare the postoperative pain of this technique to another common technique used in our clinic. Postoperative pain after one-visit root-canal treatment on teeth with vital pulps: Comparison of three different obturation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asymptomatic or symptomatic irreversible pulpitis according to AAE consensus. The diagnosis was based on clinical examinations and confirmed upon accessing the teeth.
* Consenting adults age 18 years and older
* Non-contributory medical history (ASA Class I & II)
* Included patients were given oral and written information agreed for participation and signed the informed consent

Exclusion Criteria:

* Non-consenting patients and patients below 18 years of age
* Medical history with ASA Class III & IV
* Non-restorable teeth
* Teeth with a non-vital pulp
* Periodontal probing depths were more than 4mm
* Pre-medication with antibiotics and/or analgesics 24 hours before the treatment
* Patients taking analgesics routinely for non-dental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu YH, Kushnir L, Kohli M, Karabucak B. Comparing the incidence of postoperative pain after root canal filling with warm vertical obturation with resin-based sealer and sealer-based obturation with calcium silicate-based sealer: a prospective clinical trial. Clin Oral Investig. 2021 Aug;25(8):5033-5042. doi: 10.1007/s00784-021-03814-x. Epub 2021 Feb 8. PMID 33555456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only recruited irreversible pulpitis cases that received single-visit root canal treatment.
Period: Overall Study
Arm/Group | Obturation Technique: WVT | Obturation Technique: SBT
Started | 97 | 97
Completed | 41 | 51
Not Completed | 56 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obturation Technique: WVT | Obturation Technique: SBT | Total
Number analyzed (Participants) | 41 | 51 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.4) | 46.7 (16.6) | 46.5 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 11 | 17 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: Patients were asked to rate the intensity of preoperative pain on a visual analogue scale (VAS) from 0 (no pain) to 10 (worst pain ever) before receiving root canal treatment. At the end of the visit, the patients were given a survey and asked to rate the intensity of postoperative pain (VAS 0-10) at 4 hours, 24 hours, and 48 hours after the procedure.
Time Frame: 4-, 24-, and 48-hour after receiving root canal treatment
Population: The data from all 92 survey was included for analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Obturation Technique: WVT | Obturation Technique: SBT
Number analyzed (Participants) | 41 | 51
score on a scale
  Preoperative | 4.06 [2.95 to 5.17] | 2.68 [1.90 to 3.45]
  Postoperative 4-hour | 2.41 [1.74 to 3.09] | 2.27 [1.65 to 2.94]
  Postoperative 24-hour | 1.95 [1.27 to 2.63] | 1.8 [1.14 to 2.49]
  Postoperative 48-hour | 1.15 [0.60 to 1.70] | 1.00 [0.54 to 1.46]

ADVERSE EVENTS:
Time Frame: 1.Preoperative 2. 4-, 24-, and 48-hour postoperatively
Arm/Group | Obturation Technique: WVT | Obturation Technique: SBT
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/51
Other Adverse Events (participants affected / at risk) | 0/41 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04462731/Prot_SAP_002.pdf
  • Informed Consent Form (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04462731/ICF_003.pdf